CLINICAL TRIAL: NCT00188617
Title: Phase II Study Of Single Agent Gefitinib (Iressa) In Patients With Clinical Stage I Non-Small Cell Lung Cancer (NSCLC) Proceeding To Mediastinoscopy And Surgery
Brief Title: Phase 2 Study Of Neoadjuvant Iressa Treatment In Stage 1 NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB04-0420-C; ASTRA ZENECA study D7913L00038
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: LUNG CANCER
Keywords: LUNG CANCER; IRESSA; GEFITINIB; STAGE 1A & 1B; NEOADJUVANT; PHASE 2
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: GEFITINIB — 250 mg once a day for 28 days before surgery
  Other Names: IRESSA

SUMMARY:
ELIGIBILITY

* Non-small cell lung cancer Clinical Stage 1A (T1N0M0 a tumor that is 3 cm or less in greatest dimension, surrounded by lung or visceral pleura, and without bronchoscopic evidence of invasion more proximal than the lobar bronchus (i.e., not in the main bronchus)* or 1B (T2N0M0 a tumor with any of the following features of size or extent: More than 3 cm in greatest dimension. Involves the main bronchus, 2 cm or more distal to the carina. Invades the visceral pleura. Associated with atelectasis or obstructive pneumonitis that extends to the hilar region but does not involve the entire lung).
* Must be deemed appropriate surgical candidate
* ECOG performance status £ 2
* Age ³ 18 years
* No prior chemotherapy, radiotherapy or EGFR inhibitors

PRE-TREATMENT INVESTIGATIONS

* History, physical examination, hematology, biochemistry, toxicity/baseline symptoms: within 7 days of registration
* Radiology: CT chest within 7 days of registration
* Tumor biopsy prior to treatment

TREATMENT

* Gefitinib 250 mg will be administered orally daily x 28 days

EVALUATIONS ON TREATMENT

* Physical examination (vital signs, weight, ECOG performance status) weekly x 4
* Hematology (CBC, differential): Day 1,15, 29
* Biochemistry (creatinine, electrolytes, bilirubin, alkaline phosphatase, AST/ALT, protein): Day 1,15, 29
* Radiology: CT at baseline and after day 28
* Toxicity evaluation: continuous

DURATION OF TREATMENT

* Treatment is to be discontinued in cases of serious or unacceptable toxicity, or by patient or physician request
* Otherwise duration of therapy will be a maximum of 28 days

DETAILED DESCRIPTION:
Primary and Secondary Outcomes:

* Objectives:

  * To assess the pathologic and radiological response rate after neoadjuvant Gefitinib treatment
  * To assess the toxicity of neoadjuvant Gefitinib treatment in clinical stage 1A & 1B NSCLC
* Enrollment

Treatment will be administered on an outpatient basis. Patients may be identified by thoracic surgeons, respirologists and/or interventional chest radiologists for study participation upon clinical and radiographic assessment.

**Diagnostic biopsy, Pretreatment Investigations

If patients have already had a core or FNA biopsy before referral, this material will be sought from the original pathologist for review and inclusion in the study with appropriate consent sought. If a patient does not have a biopsy upon presentation to the thoracic surgeon, and consents to inclusion in the trial, baseline non-invasive assessment will be carried out before a percutaneous biopsy will be mandated as part of entry into the study. After non-invasive staging, patients will be subject to biopsy. In collaboration with pathology, an immediate diagnosis will be made at the time of fine needle aspiration biopsy (or bronchoscopy). After a pathologic diagnosis of cancer is confirmed, subjects will be invited to have additional biopsies will be performed to obtain material for correlative studies, assuming no complications or technical difficulties have arisen. These studies will be done in collaboration with thoracic interventional radiologists from Diagnostic Imaging, who supervises the lung fine needle aspirates and biopsies.

All patients will undergo pre-study assessments for symptoms, performance status, radiographic assessment and blood tests (complete blood count, electrolytes, liver and renal function tests). Assessment of response will occur after the 4-week treatment period. Toxicity will be assessed continuously, with patient assessment weekly on treatment, repeat blood tests at 2 weeks and imaging of measurable disease at 4 weeks. All subjects will be invited to have their initial diagnostic biopsy and subsequent surgical tumor specimen examined as part of the laboratory correlate component of the study. Patients will be considered evaluable for pharmacodynamic assessment if they complete at least 21 of the planned 28 days of therapy.

Once competed, oral Gefitinib will be administered at a dose of 250 mg (1 pill) daily for 28 days prior to the planned mediastinoscopy. Patients may take the pill either with or without food, and are encouraged to take the medication at approximately the same time each day. If the patient forgets to take a dose, they should take the last missed dose as soon as they remember, as long as it is at least 12 hours before the next dose is due. If patient vomits after taking the dose, the dose may be retaken if the tablet is seen in the emesis. The last dose of Gefitinib will be administered not less than 48 hours prior to mediastinoscopy or surgery.

If the mediastinoscopy reveals the presence of Stage III disease, the patient's mediastinoscopy samples may still be analysed as part of the correlative study. Patients will be followed for 90 days or as long as required after the last dose of Gefitinib to ensure resolution of any Gefitinib-related toxicities. However these patients will be offered standard therapy for stage III disease off of study protocol, for example a combination of chemotherapy, radiation plus or minus surgical resection. If these patients do proceed to thoracotomy post-chemotherapy and/or radiotherapy, their resection specimen will not be eligible for this correlative protocol.

**Duration of Therapy and Follow-up

As outlined above, patients will be treated for 28 days before surgery and will also be followed for 90 days post-operatively after thoracotomy to ensure the recovery from surgery. Accrual is estimated at 2 patients per month, for 18 to 24 months, based on accrual rates to other thoracic surgical studies at UHN. Study duration is planned from August 2004 to June 2006.

All patients will be followed in the current standard of care at University Health Network. That is, clinic visits with chest x-ray every 3 months for 2 years, every 6 months in the third year, and annually thereafter. Recorded information will only include vital status and presence or absence of disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven non-small cell lung carcinoma (NSCLC) or a lung nodule seen on CT imaging and a high-clinical suspicion of NSCLC
* Clinical Stage 1A (T1N0M0 a tumor that is 3 cm or less in greatest dimension, surrounded by lung or visceral pleura, and without bronchoscopic evidence of invasion more proximal than the lobar bronchus (i.e., not in the main bronchus)
* or 1B (T2N0M0 a tumor with any of the following features of size or extent: More than 3 cm in greatest dimension. Involves the main bronchus, 2 cm or more distal to the carina. Invades the visceral pleura. Associated with atelectasis or obstructive pneumonitis that extends to the hilar region but does not involve the entire lung).

  * Must be deemed appropriate surgical candidate
  * ECOG performance status £ 2
  * Age ³ 18 years
  * No prior chemotherapy, radiotherapy or EGFR inhibitors
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have received prior anticancer treatment with chemotherapy, radiotherapy or EGFR inhibitor therapy;
* Patients who have had a previous diagnosis of cancer, are excluded except if have been adequately treated for non-melanoma skin cancer or carcinoma in situ of the cervix are eligible irrespective of when that treatment was given.
* Patients may not be receiving any other investigational or anticancer agents while on study;
* History of allergic reactions to Gefitinib or erlotinib
* Pre-existing diarrhea ³ NCI CTC Grade 2
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure or evidence of cardiac dysfunction, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease, poorly controlled diabetes mellitus, clinically significant or untreated ophthalmologic (e.g. Sjogrens etc.) or gastrointestinal conditions (e.g. Crohns disease, ulcerative colitis) or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women because of the unknown effects of Gefitinib on the human fetus.
* HIV-positive patients on active treatment
* Active malignancy at any other site including combined small cell and non-small cell carcinomas or a pulmonary carcinoid tumor.
* Taking drugs that induce CYP3A4 enzymes, patients with ongoing use of phenytoin, rifampicin, carbamazepine, barbiturates, rifampicin, or St John's Wort are excluded.
* Incomplete healing from previous surgery.
* Use of any agent that decreases gastric pH, including proton pump inhibitors, Histamine-2 receptor blockers or sodium bicarbonate. Use of calcium or magnesium based elixirs are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
· To assess the pathologic and radiological response rate after neoadjuvant Gefitinib treatment | before starting drug and after 28 days of treatment

SECONDARY OUTCOMES:
· To assess the toxicity of neoadjuvant Gefitinib treatment in clinical stage 1A & 1B NSCLC | at baseline, 2weeks into treatment at 4weeks and 30 days after stopping drug

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waddell, MD FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada